CLINICAL TRIAL: NCT01491841
Title: Phase I/II Study of the Combination of Bendamustine, Rituximab and Pixantrone in Patients With Relapsed/Refractory B Cell Non-Hodgkin's Lymphoma
Brief Title: IIT CTI Bendamustine, Rituximab, Pixantrone in Relapsed/Refractory B Cell Non-Hodgkin's Lymphoma
Acronym: BRP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anne Beaven, MD (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor-Investigator, Anne Beaven, MD, Assist Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030834
Record Dates: First submitted 2011-11-14; First posted 2011-12-14 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; Rituximab; pixantrone; pegfilgrastim

STUDY DESIGN:
Intervention Model Description: Dose Escalation, 3+3 design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Pixantrone, 55mg/m^2 (Experimental): Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 55mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Interventions: Drug: Bendamustine + Rituximab + Pixantrone; Drug: Pegfilgrastim
- Phase 1: Pixantrone, 85mg/m^2 (Experimental): Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 85mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Interventions: Drug: Bendamustine + Rituximab + Pixantrone; Drug: Pegfilgrastim
- Phase 1: Pixantrone, 115mg/m^2 (Experimental): Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 115mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Interventions: Drug: Bendamustine + Rituximab + Pixantrone; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Bendamustine + Rituximab + Pixantrone — Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
  Other Names: BRP; BuRP
Drug: Pegfilgrastim — 6mg administered on Day 2 of each 21 day cycle

SUMMARY:
This is a phase I trial of the combination of bendamustine, rituximab and pixantrone in patients with relapsed/refractory B cell non-Hodgkin lymphoma. A standard 3+3 design will be used to determine the maximum tolerated dose (MTD) of the combination. A static dose of bendamustine and rituximab will be used and the dose of pixantrone will be escalated in each cohort. Pixantrone will be dosed on a 21 day cycle at 55mg/m2, 85mg/m2, and 115mg/m2 in sequential cohorts dependent on acceptable toxicity profile at each dose level. MTD will be determined based on DLTs that occur during the first 2 cycles of the drug combination.

Phase II did not proceed as planned due to withdrawal of pixantrone from the US.

DETAILED DESCRIPTION:
This is a phase I trial utilizing a traditional 3+3 design to evaluate maximum tolerated dose (MTD) and optimal dose schedule of pixantrone in combination with bendamustine (120mg/m2 on day 1 of each 21 day cycle) and rituximab (375mg/m2 on day 1 of each 21 day cycle). No patients will be entered on an escalated dosage level until at least 3 patients have been treated at the previous level and assessed for a dose limiting toxicity. Dose levels will be escalated in cohorts of 3 patients as long as no drug-related DLT occurs in the first 2 cycles. If one patient is observed to suffer a DLT, this cohort will be expanded to include at least 6 patients total. If less than 2 patients in the expanded cohort of 6 patients experience a DLT, dose escalation will resume. If 2 of 6 patients enrolled at the same dose level experience a DLT, the MTD has been exceeded, and the dose escalation will cease. The next lower dose will be considered the MTD. If any patient withdraws from the study prior to completing 2 cycles for reasons other than a DLT then that patient will be replaced in order to determine the MTD.

If dose limiting toxicity is observed at the initial dose level in 2 patients, the MTD has been exceeded and the starting dose level will be reduced to 25mg/m2. If 1 patient experiences a DLT in the -1 dose range, the cohort will be expanded to at least 6 patients. If a second patient experiences a DLT at the -1 dose level, the trial will be closed.

For part 1, those who have a confirmed diagnosis of relapsed/refractory B cell non-Hodgkin's lymphoma of any subtype will be considered eligible for enrollment. Each cycle will be 21 days. Subjects will be assessed for DLTs during the first 2 cycles of study drug. They will be assessed for response after cycle 2. Patients not experiencing a DLT during the first 2 cycles and who have stable disease or better may continue to receive up to 6 cycles of treatment with the triplet combination. If any patient withdraws from the study prior to completing 2 cycles for reasons other than a DLT then that patient will be replaced in order to determine the MTD.

Phase II did not proceed as planned due to withdrawal of pixantrone from the US.

ELIGIBILITY:
Inclusion Criteria:

1. Part I: Subjects must have relapsed or refractory B cell NHL;
2. Part II: Subjects must have relapsed or refractory aggressive B cell NHL including follicular lymphoma (FL) grade 3, Diffuse Large B Cell Lymphoma (DLBCL), transformed NHL, mantle cell lymphoma (MCL), or other aggressive B cell NHL histology as per the WHO 2008 criteria;
3. Refractory disease (defined as persistence of evaluable disease after therapy) or relapsed disease following at least one prior treatment regimen that should include autologous stem cell transplant unless a patient was not eligible or refused prior transplant;
4. Age ≥ 18 years old;
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2;
6. Subjects must have measurable or evaluable disease based on physical exam and/or radiographs (CT, MRI, PET) or bone marrow involvement;
7. Female subject is either post-menopausal or surgically sterilized;
8. Laboratory Values:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; lower levels accepted if due to marrow involvement by lymphoma
   * Platelets ≥ 75,000/mcl; lower levels accepted if due to marrow involvement by lymphoma
   * Total bilirubin ≤ 1.5 X institutional upper limit of normal; ≤ 3.0 ULN accepted in subjects with Gilbert's Syndrome
   * AST/ALT ≤ 1.5 X institutional upper limit of normal. Subjects with known liver involvement by lymphoma: AST/ALT ≤ 2 X institutional upper limit of normal
   * Serum creatinine < 1.5 X institutional upper limit of normal
9. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed

Exclusion Criteria:

1. No chemotherapy, radiation, biologics or immunotherapy within 2 weeks prior to registration (6 weeks if last received BCNU or mitomycin C).
2. No radioimmunotherapy within 2 months prior to registration.
3. Subjects receiving chronic, systemic treatment with corticosteroids equivalent to > 20mg of prednisone per day. Subjects receiving replacement for adrenal insufficiency will be allowed on the study. Topical or inhaled corticosteroids are allowed.
4. Subjects with a history of another primary malignancy ≤ 3 years ago, with the exception of inactive basal, squamous cell carcinoma of the skin or superficial melanoma only requiring excision, prostate cancer with a PSA that has not increased for at least 3 months, carcinoma in situ of the cervix.
5. Major surgery ≤ 4 weeks prior to registration. Minor surgery ≤ 2 weeks prior to registration. Insertion of a vascular access device is not considered major or minor surgery. Subjects must have recovered from all surgery related toxicities to ≤ grade 1 or to baseline if subject started with > grade 1 toxicity, not otherwise violating the above inclusion criteria.
6. Subjects who have received investigational drugs ≤ 4 weeks prior to registration.
7. Impaired Cardiac Function:

   * QTc > 480 on screening ECG.
   * Previous history of angina pectoris or acute MI within 6 months
   * Congestive heart failure (New York Heart Association functional classification III-IV) or baseline MUGA/ECHO shows estimated LVEF < 45%
   * Any history of torsade de pointes, ventricular fibrillation, uncontrolled ventricular tachycardia, or uncontrolled atrial fibrillation.
8. Female patients who are pregnant or breastfeeding
9. Patients with history of untreated hepatitis B or who are known carriers of hepatitis B will be excluded from this trial. All subjects will be screened prior to study entry.
10. Concurrent use of other anti-cancer agents or anti-cancer treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened November 1, 2011 and closed to accrual September 22, 2016. Subjects were recruited through the Hematology Clinic at Duke University Medical Center.
Groups:
- Bendamustine + Rituximab + Pixantrone: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, variable dosing depending on the cohort and MTD (maximum tolerated dose); to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Bendamustine + Rituximab + Pixantrone: Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
Period: Overall Study
Arm/Group | Bendamustine + Rituximab + Pixantrone
Started | 33
Completed | 22
Not Completed | 11
Not completed — Screen Failure | 10
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Bendamustine + Rituximab + Pixantrone: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, variable dosing depending on the cohort and MTD; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Bendamustine + Rituximab + Pixantrone: Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
Arm/Group | Bendamustine + Rituximab + Pixantrone
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Dose-limiting toxicity (DLT) assessments were performed weekly during cycles 1 and 2. A DLT was defined as any grade 3 non-hematologic toxicity that lasted longer than 48 hours, despite proper supportive care, any grade 4 non-hematologic toxicity, or any grade 3 or 4 hematologic toxicity lasting longer than 7 days. Alopecia and febrile neutropenia were not considered DLTs. Any NCI CTC (National Cancer Institute Common Terminology Criteria) v4.03 grade 5 (death) toxicity was considered a DLT. Dose Limiting Toxicities were used as the assessment criteria to determine the Maximum Tolerated Dose (MTD). MTD is presented.
Time Frame: 4 years
Population: Over the course of 4 years, dose escalation was performed in 3 cohorts. Cohort 1 (Phase 1: Pixantrone, 55mg/m^2) enrolled 7 people; Cohort 2 (Phase 1: Pixantrone, 85mg/m^2) enrolled 7 people; Cohort 3 (Phase 1: Pixantrone, 115 mg/m^2) enrolled 7 people.
Measure: Number; unit: milligrams per meter squared
Groups:
- Bendamustine + Rituximab + Pixantrone + Pegfilgrastim: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, variable dosing depending on the cohort and MTD; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Bendamustine + Rituximab + Pixantrone: Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
Arm/Group | Bendamustine + Rituximab + Pixantrone + Pegfilgrastim
Number analyzed (Participants) | 21
milligrams per meter squared | 115

2. Secondary Outcome: Overall Response
Description: Partial response and complete response evaluated using a modified version of the revised response criteria for malignant lymphoma by Cheson et al
  Complete Response (CR) • Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present prior to therapy.
  Complete Response Unconfirmed (CRu) meets the CR criteria, but with one or more of the following:
  * A residual node > 1.5 cm in greatest transverse diameter that has regressed >75% in the sum of the product of the diameters (SPD). Individual nodes that were previously confluent must have regressed >75% in their SPD compared with the size of the original mass.
  * Indeterminate bone marrow (increased number or size of aggregates without cytologic or architectural atypia by immunohistochemistry or flow cytometry).
  Partial Response (PR)
  • A decrease of ≥ 50% in the SPD of up to six of the largest dominant nodes or nodal masses.
Time Frame: up to 220 days
Population: Subjects who received at least 2 cycles of study drug were included. Data from the single patient enrolled in the phase 2 portion of the trial was included with the phase I pixantrone 115mg/m2 group because the phase 2 patient also received the 115mg/m2 dose and the combined data seems more meaningful than presenting data for 1 patient separately.
Measure: Count of Participants; unit: Participants
Groups:
- Pixantrone, 55mg/m^2: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 55mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Bendamustine + Rituximab + Pixantrone: Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
- Pixantrone, 85mg/m^2: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 85mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Bendamustine + Rituximab + Pixantrone: Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
- Pixantrone, 115mg/m^2: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 115mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
  Bendamustine + Rituximab + Pixantrone: Dose escalation of pixantrone (55mg/m2, 85mg/m2 and 115mg/m2) in combination with static dose bendamustine (120mg/m2 on Day 1 of each 21 day) and rituximab (375mg/m2 on Day 1 of each 21 day cycle).
Arm/Group | Pixantrone, 55mg/m^2 | Pixantrone, 85mg/m^2 | Pixantrone, 115mg/m^2
Number analyzed (Participants) | 4 | 3 | 7
Participants | 2 | 2 | 5

3. Secondary Outcome: Progression Free Survival
Time Frame: From day 1 of treatment to disease progression, death or 5 years, whichever comes first
Population: Groups combined to include all subjects who completed the study. This analysis was originally planned for Phase 2; there was no intent to compare dose levels in Phase 1 because there would be insufficient power to make meaningful comparisons.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab + Pixantrone + Pegfilgrastim
Number analyzed (Participants) | 22
months | 3.9 [1.3 to 6.9]

4. Secondary Outcome: Toxicity
Description: Dose limiting toxicities plus % of patients with a clinically significant change in left ventricular ejection fraction.
Time Frame: 30 days post last dose of study drug
Population: Phase 1 subjects who received study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Pixantrone, 55mg/m^2 | Phase 1: Pixantrone, 85mg/m^2 | Phase 1: Pixantrone, 115mg/m^2
Number analyzed (Participants) | 7 | 7 | 7
Participants
  Dose-Limiting Toxicity | 1 | 1 | 1
  Left Ventricular Ejection Fraction | 1 | 0 | 0
  Other Adverse Events | 6 | 6 | 6

5. Secondary Outcome: Overall Survival
Time Frame: from day 1 of treatment to death
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine + Rituximab + Pixantrone + Pegfilgrastim
Number analyzed (Participants) | 22
months | 7.9 [4.2 to 15.4]

ADVERSE EVENTS:
Time Frame: Up to 220 days
Description: Subjects who received at least 2 cycles of study drug were included. Data from the single patient enrolled in the phase 2 portion of the trial was included with the phase I pixantrone 115mg/m2 group because the phase 2 patient also received the 115mg/m2 dose and the combined data seems more meaningful than presenting data for 1 patient separately.
Groups:
- Pixantrone, 55mg/m^2: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 55mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
- Pixantrone, 85mg/m^2: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 85mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
- Pixantrone, 115mg/m^2: Bendamustine, 120mg/m2; administered first on Day 1 of each cycle. Rituximab, 375mg/m2; administered second on Day 1 of each cycle. Pixantrone, 115mg/m2; to be administered last, 4-6 hours after bendamustine, on Day 1 of each cycle Pegfilgrastim, 6mg; administered on Day 2 of each cycle
Arm/Group | Pixantrone, 55mg/m^2 | Pixantrone, 85mg/m^2 | Pixantrone, 115mg/m^2
All-Cause Mortality (participants affected / at risk) | 6/7 | 7/7 | 8/8
Serious Adverse Events (participants affected / at risk) | 3/7 | 0/7 | 2/8
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pixantrone, 55mg/m^2 (N=7) | Pixantrone, 85mg/m^2 (N=7) | Pixantrone, 115mg/m^2 (N=8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pixantrone, 55mg/m^2 (N=7) | Pixantrone, 85mg/m^2 (N=7) | Pixantrone, 115mg/m^2 (N=8)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 4
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 4
Edema limbs (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 5 | 2 | 6
Fever (General disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Gum infection (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3
Creatinine increased (Investigations) | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 4
Platelet count decreased (Investigations) | 2 | 0 | 5
Urine output decreased (Investigations) | 0 | 0 | 1
Weight loss (Investigations) | 2 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes